CLINICAL TRIAL: NCT06562244
Title: A Family-focused Intervention Program to Foster Adolescent Mental Health and Well-being: Protocol for a Multi-country Cluster Randomized Factorial Trial (FLOURISH Phase 2)
Brief Title: Family-Focused Adolescent &Amp; Lifelong Health Promotion Optimization Trial
Acronym: FLOURISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Klagenfurt (Other)
Collaborators: Institute for Marriage, Family and Systemic Practice - ALTERNATIVA (Other); Cardiff University (Other); Association for Systematic Therapy Education Center (Unknown); Medical University of Vienna (Other); University Jaume I Castellon (Unknown); Bielefeld University (Other); Health for Youth Association, Moldova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1010955282
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Adolescent - Emotional Problem; Parent-Child Relations; Family Functioning; Well-Being, Psychological
Keywords: Multiphase Optimization Strategy (MOST); Family-based intervention; Adolescents; Mental health; Randomized trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- HAT On, Peer Support On, High Engagement (Experimental): HAT component: On - Two interactive sessions using UNICEF's Helping Adolescents Thrive comics, covering recognizing emotions, stress management, conflict resolution, and relationship building.
  Peer Support: On - Half-day workshop from UNICEF's "I Support My Friends" program, teaching adolescents to identify distress in peers, develop listening skills, and seek additional support.
  Engagement booster: High - Includes refreshments, certificates, and vouchers (10 EUR for adolescents, 5 EUR for caregivers).
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH); Behavioral: Helping Adolescents Thrive comics; Behavioral: I Support My Friends
- HAT On, Peer Support Off, High Engagement (Experimental): HAT component: On - Two interactive sessions using UNICEF's Helping Adolescents Thrive comics, covering recognizing emotions, stress management, conflict resolution, and relationship building.
  Peer Support: Off
  Engagement booster: High - Includes refreshments, certificates, and vouchers (10 EUR for adolescents, 5 EUR for caregivers).
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH); Behavioral: Helping Adolescents Thrive comics
- HAT On, Peer Support On, Low Engagement (Experimental): HAT component: On - Two interactive sessions using UNICEF's Helping Adolescents Thrive comics, covering recognizing emotions, stress management, conflict resolution, and relationship building.
  Peer Support: On - Half-day workshop from UNICEF's "I Support My Friends" program, teaching adolescents to identify distress in peers, develop listening skills, and seek additional support.
  Engagement booster: Low - Refreshments and certificates.
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH); Behavioral: Helping Adolescents Thrive comics; Behavioral: I Support My Friends
- HAT On, Peer Support Off, Low Engagement (Experimental): HAT component: On - Two interactive sessions using UNICEF's Helping Adolescents Thrive comics, covering recognizing emotions, stress management, conflict resolution, and relationship building.
  Peer Support: Off
  Engagement booster: Low - Refreshments and certificates.
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH); Behavioral: Helping Adolescents Thrive comics
- HAT Off, Peer Support On, High Engagement (Experimental): HAT component: Off
  Peer Support: On - Half-day workshop from UNICEF's "I Support My Friends" program, teaching adolescents to identify distress in peers, develop listening skills, and seek additional support.
  Engagement booster: High - Includes refreshments, certificates, and vouchers (10 EUR for adolescents, 5 EUR for caregivers).
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH); Behavioral: I Support My Friends
- HAT Off, Peer Support Off, High Engagement (Experimental): HAT component: Off
  Peer Support: Off
  Engagement booster: High - Includes refreshments, certificates, and vouchers (10 EUR for adolescents, 5 EUR for caregivers).
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH)
- HAT Off, Peer Support On, Low Engagement (Experimental): HAT component: Off
  Peer Support: On - Half-day workshop from UNICEF's "I Support My Friends" program, teaching adolescents to identify distress in peers, develop listening skills, and seek additional support.
  Engagement booster: Low - Refreshments and certificates.
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH); Behavioral: I Support My Friends
- HAT Off, Peer Support Off, Low Engagement (Experimental): HAT component: Off
  Peer Support: Off
  Engagement booster: Low - Refreshments and certificates
  Interventions: Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH)

INTERVENTIONS:
Behavioral: Parenting for Lifelong Health for Parents and Teens (PLH) — The PLH program is the core intervention and will be delivered over 6 sessions with adolescents and caregivers, focusing on building positive parent-child relationships, problem-solving skills, stress management, effective limit-setting, and emotional regulation. There will also be a pre-program visit with the facilitator and families prior to the group sessions. Sessions will include both separate and joint activities between adolescents and caregivers. Engagement boosters will be provided during the PLH sessions and are part of the PLH intervention.
Behavioral: Helping Adolescents Thrive comics — UNICEF's Helping Adolescents Thrive (HAT) comics will be used to guide adolescents through content on improving relationships, handling conflict, understanding emotions, and problem solving. These sessions will be group-based and cover the content in the HAT manual with the adolescents in an interactive format.
  Arms: HAT On, Peer Support Off, High Engagement; HAT On, Peer Support Off, Low Engagement; HAT On, Peer Support On, High Engagement; HAT On, Peer Support On, Low Engagement
Behavioral: I Support My Friends — An adapted version of UNICEF's "I Support My Friends" program will be provided to adolescents by a facilitator in a group-based workshop format over the course of 1 day.
  Arms: HAT Off, Peer Support On, High Engagement; HAT Off, Peer Support On, Low Engagement; HAT On, Peer Support On, High Engagement; HAT On, Peer Support On, Low Engagement

SUMMARY:
The aim of this study is to conduct a multi-country, cluster-randomized factorial trial to optimize the Parenting for Lifelong Health (PLH) for Parents and Teens program in Moldova and North Macedonia. Specifically, this trial will evaluate the effectiveness and cost consequences of three additional intervention components: UNICEF's Helping Adolescents Thrive comics, adolescent peer support based on UNICEF's I Support My Friends intervention, and engagement boosters.

ALTERNATIVA will deliver the program in North Macedonia and Health for Youth Association in the Republic of Moldova.

This trial is implemented according to the Multiphase Optimization Strategy (MOST). MOST involves three phases. The preparation phase involves adapting and piloting the intervention (Phase 1). The optimization phase involves a factorial trial (Phase 2). Finally, the evaluation phase involves conducting a randomized controlled trial to assess the optimized intervention's effectiveness and cost-effectiveness (Phase 3). A Phase 2 factorial trial is the focus of this registration.

DETAILED DESCRIPTION:
Adolescent mental health is a significant global concern, especially in low- and middle-income countries (LMICs) like North Macedonia and Moldova. Adolescents in LMICs face numerous challenges, including socio-economic stressors, adverse childhood experiences, and limited access to mental health services. Parenting interventions are one approach to reduce risk for poor adolescent mental health outcomes and family maltreatment. Systematic optimization of parenting programs is essential for enhancing scalability and sustainability in low-resource settings.

Building on prior research, the "Family-Focused Adolescent & Lifelong Health Promotion" (FLOURISH) project aims to adapt, optimize, and evaluate a parenting intervention for adolescents aged 10-14 and their caregivers in North Macedonia and Moldova. The project focuses on improving adolescent mental health and well-being in both teens and caregivers, and it is implemented according to the Multiphase Optimization Strategy (MOST) framework. Phase 1 of the project assessed the feasibility of the adapted parenting intervention, which included three components to enhance participation, retention, and effectiveness. The three components were UNICEF's Helping Adolescents Thrive (HAT) comics, peer support, and engagement boosters.

This protocol describes the optimization (Phase 2) of the adapted FLOURISH intervention package which will assess the effectiveness and costs of HAT, adolescent peer support, and the engagement boosters, as well as their combinations. The factorial experiment will consist of eight conditions, stratified by country, with each condition reflecting a unique combination of the three components. The results of this study will be used to select the optimized intervention package which will be tested in a randomized trial in the next phase of the FLOURISH project (Phase 3).

ELIGIBILITY:
Inclusion Criteria:

For Caregivers:

Must be 18 years or older at the baseline assessment. Must be the primary caregiver of an adolescent aged 10-14 who has resided in the same household for at least four nights a week in the past month.

Must be able to speak at least one of the local languages in which the program will be offered (Romanian, Macedonian).

Must agree to participate in the program. Must provide consent for both themselves and their child to participate in the study.

For Adolescents:

Must be aged 10-14 at the baseline assessment. Must assent to participate in the study. Must have caregiver consent to participate in the study.

Exclusion Criteria:

No formal exclusion criteria have been established for the FLOURISH project. However, during the project introduction, the research team will guide participants through a consent form that asks whether they are currently experiencing acute distress or a mental or physical health condition that could interfere with their participation. The decision will be made by the potential participant. If the participant decides they are unable to take part due to acute health issues, the research team will follow up and provide referrals to other services.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 640 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in levels of caregiver-reported emotional problems in adolescents: Child Behavior Checklist (CBCL) 6-18, "internalizing subscale" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CBCL is an instrument from the Achenbach System of Empirically Based Assessment (ASEBA). Each problem item is rated 0=not true, 1=somewhat or sometimes true, and 2=very true or often true. Standardized scores can be computed with higher scores indicating more problems.
Change in levels of social support in adolescents: Medical Outcome Study Social Support Survey (MOS-SSS), "emotional support subscale", and Kidscreen-52, "peer and social support subscale" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The MOS-SSS includes 18 items with a response range from 1 (none of the time) to 5 (all of the time). The emotional support scale comprises 8 items. The Kidscreen-52, peers and social support subscale, includes 6 items with a response range from 1 (never) to 5 (always). This subscale assesses the quality of the child's relationships with peers and the support they receive from their social network.
Change in levels of family functioning in caregivers: Family Assessment Device (FAD), subscale "general functioning" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The general functioning subscale is one of the dimensions of the FAD and will be completed by caregivers. This scale has also been used as a single indicator to assess family functioning. The general functioning scale is made up of 12 items with six items that reflect healthy family functioning and the other six items reflecting unhealthy functioning. Scoring is on a 4-point scale (from 1 for strongly agree to 4 for strongly disagree) with the scoring for the negatively worded items reversed.
Attendance rate | During the implementation of the intervention (6 - 8 weeks)
  Attendance will be assessed as the percentage of group PLH sessions attended out of 6 (individual attendance for adolescents and caregivers)

SECONDARY OUTCOMES:
Change in levels of family communication in adolescents: Child-Parent Communication Apprehension scale (CPA-YA), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CPA-YA measures parent-child communication apprehension and will be completed by adolescents. The tools consists of 12 items with responses being scored using a 5-point Likert-type scale, from 1 (strongly disagree) to 5 (strongly agree).
Change in frequency of parenting practices: Alabama Parenting Questionnaire-APQ, subscale "involved parenting" and "positive parenting" (parent- and child-report), and subscale "corporal punishment" (parent-report) | Pre-Post (approximately 6 - 8 weeks after pre-assessment)
  Parenting practices will be assessed with the child- and parent-report version of the Alabama Parenting Questionnaire (APQ). The APQ is a self-report measure of parenting behaviors designed to assess the parenting practices most related to disruptive behaviors of children. The APQ subscales may be rated by parents and children (caregiver-report and child-report) using a 5-point scale ranging from 1 (never) to 5 (always).
Change in levels of loneliness in adolescents: UCLA-8 Loneliness scale, total score | Pre-Post (approximately 6 - 8 weeks after pre-assessment)
  The UCLA-8 is brief 8-item version developed specifically for use with adolescents. Items are scored on 4-point scale.
Change in levels of social support in adolescents: Medical Outcome Study Social Support Survey (MOS-SSS), "affectionate subscale" | Pre-Post (approximately 6 - 8 weeks after pre-assessment)
  The MOS-SSS includes 18 items with a response range from 1 (none of the time) to 5 (all of the time). The affectionate support subscale comprises 3 items.
Change in levels of well-being in adolescents and caregivers: World Health Organization-Five Well-Being Index (WHO-5), total score | Pre-Post (approximately 6 - 8 weeks after pre-assessment)
  The WHO-5 is a short, positively worded instrument designed to assess the level of emotional well-being over 14 days. Respondents are asked to rate how well each of the 5 statements applies to them when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). Therefore, the raw score theoretically ranges from 0 (absence of well-being) to 25 (maximal well-being).
Change in levels of psychological distress in caregivers: Patient Health Questionnaire - 9 (PHQ-9), total score | Pre-Post (approximately 6 - 8 weeks after pre-assessment)
  The PHQ-9 is a 9-item self-report questionnaire used as a continuous measure to assess depressive symptom severity. Response options on the items range from 'not at all' (0 points) to 'nearly every day' (3 points).
Change in levels of parental stress in caregivers: Parental Stress Scale (PSS), total score | Pre-Post (approximately 6 - 8 weeks after pre-assessment)
  The PSS is an 18-item self-report questionnaire. Items are rated on a 5-point Likert scale (1 = Strongly disagree, 2 = Disagree, 3 = Undecided, 4 = Agree, 5 = Strongly agree) and scores range from 18 to 90, with higher values indicating greater levels of parental stress.
Change in levels of emotional problems in adolescents: Revised Child Anxiety and Depression Scales (RCADS), total score, "depression and anxiety subscales" | Pre-Post (approximately 6 - 8 weeks after pre-assessment)
  The RCADS requires respondents to rate how often each item applies to them. Items are scored 0-3 corresponding to ''never,'' ''sometimes,'' ''often,'' and ''always''.
Change in levels of loneliness in caregivers: Revised UCLA Loneliness scale (RULS-6), total score | Pre-Post (approximately 6 - 8 weeks after pre-assessment)
  The RULS-6 was developed as a short 6-item version suitable for use among adults.
Change in levels of caregiver-reported behavior problems in adolescents: Child Behavior Checklist (CBCL) 6-18, parent-report, subscales "rule-breaking and aggressive behavior, externalizing behavior" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CBCL is an instrument from the Achenbach System of Empirically Based Assessment (ASEBA). The CBCL is a widely used instrument for assessing child behavioral and emotional symptoms.
  Each problem item is rated 0=not true, 1=somewhat or sometimes true, and 2=very true or often true. Standardized scores can be computed with higher scores indicating more problems.
Change in levels of social support in caregivers: Medical Outcome Study Social Support Survey (MOS-SSS), "emotional and affectionate subscales" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The MOS-SSS includes 18 items with a response range from 1 (none of the time) to 5 (all of the time). The emotional and affectionate support scales comprise 11 items.
Change in levels of family functioning in caregivers: Family Assessment Device (FAD), "problem solving and communication subscales" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The FAD measures changes in family functioning among caregivers. The problem solving subscale includes 6 items that assess the family's ability to resolve problems effectively. The communication subscale comprises 9 items that evaluate the clarity and directness of information exchange within the family. Responses for both subscales range from 1 (strongly agree) to 4 (strongly disagree).
Change in levels of emotional problems in adolescents: Pediatric Symptom Checklist (PSC), adolescent and caregiver report, total score, "internalizing, externalizing and attention subscales" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The PSC includes 17 items with a response range from 0 (never) to 2 (often), assessing emotional problems in adolescents. The checklist includes subscales for internalizing problems, externalizing problems, and attention problems.
Change in adolescent socio-emotional skills: Social Emotional Abilities and Learning (SEAL) Tool, "emotional regulation, stress management, problem-solving, interpersonal skills, and self-esteem subscales" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The subscales include 11 items with responses ranging from "yes" to "no" and "maybe".
Change in adolescent health-related quality of life: EQ-5D-Y-3L | Pre-assessment and 6 - 8 weeks after pre-assessment
  The EQ-5D-Y-3L is a standardized instrument developed to measure health-related quality of life, particularly in younger populations. It includes five distinct dimensions that assess various aspects of the respondent's health. The tool includes 5 items, each with 3 response levels: no problems, some problems, and severe problems. Additionally, it includes a visual analogue scale (VAS) where respondents rate their overall health on a scale from 0 to 100, with 0 representing the worst imaginable health and 100 representing the best imaginable health.
Change in caregiver health-related quality of life: EQ-5D-5L | Pre-assessment and 6 - 8 weeks after pre-assessment
  The EQ-5D-5L is a standardized instrument developed to measure health-related quality of life. It includes five distinct dimensions that assess various aspects of the respondent's health. The tool includes 5 items, each with 5 response levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Additionally, it includes a visual analogue scale (VAS) where respondents rate their overall health on a scale from 0 to 100, with 0 representing the worst imaginable health and 100 representing the best imaginable health.
Change in caregiver capabilities: Oxford CAPabilities questionnaire - Mental Health (OxCAP-MH) | Pre-assessment and 6 - 8 weeks after pre-assessment
  The OxCAP-MH includes 16 items assessing various dimensions of well-being and functioning, such as social participation, emotional stability, and access to resources. Response options include a 5-point Likert scale.
Change in caregiver resource use: PECUNIA Resource Use Measurement (PECUNIA RUM) | Pre-assessment and 6 - 8 weeks after pre-assessment
  The PECUNIA RUM assesses resource use through different modules such as residential care, non-residential health and social care, informal help and work.
Change in caregiver-reported resource use in adolescents: PECUNIA Resource Use Measurement (PECUNIA RUM) proxy for adolescents | Pre-assessment and 6 - 8 weeks after pre-assessment
  The PECUNIA RUM proxy for adolescents assesses resource use by adolescents through caregiver report, and cover modules such as residential care, non-residential health and social care, and education.

OTHER OUTCOMES:
Adolescent healthy weight: BMI; adolescent and caregiver reports | Pre-assessment and 6 - 8 weeks after pre-assessment
  Adolescent healthy weight will be assessed with caregiver and adolescents report on the adolescent's mass in kilograms and height in meters. This is not expected to change as a result of the intervention, but is assessed for sample description.
Caregiver alcohol use: The Alcohol Use Disorder Identification Test (AUDIT), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The AUDIT contains 10 questions concerning alcohol consumption, drinking behaviors, and alcohol-related problems. It is scored from 0 to 4 for each question, resulting in a total score ranging from 0 to 40.
Post-traumatic stress in caregivers: PTSD checklist for DSM-5 (PCL-5), short form, total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The 4-item version of the PCL-5 is a short form of the original PCL-5 consisting of 20 items. These are rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely), with higher scores indicating greater symptom severity. This tool is particularly useful for screening purposes and includes Criterion A, which refers to exposure to actual or threatened death, serious injury, or sexual violence, as a critical aspect of assessing PTSD symptoms. The tool will be completed by caregivers.
Posttraumatic stress in adolescents: Children's Revised Impact of Event Scale (CRIES), total score, "intrusion and avoidance subscales" | Pre-assessment and 6 - 8 weeks after pre-assessment
  The CRIES is organized into two dimensions-intrusion (4 items) and avoidance (4 items) and a total score. The items are scored on a four-point scale: "not at all" receives 0 scores, "rarely" sums 1 point, "sometimes" adds 3 points, and "often" computes 5 points. This tool will be completed by adolescents.
Well-being among intervention staff: World Health Organization-Five Well-Being Index (WHO-5), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The WHO-5 is a short, positively worded instrument designed to assess the level of emotional well-being over 14 days. Respondents are asked to rate how well each of the 5 statements applies to them when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). Therefore, the raw score theoretically ranges from 0 (absence of well-being) to 25 (maximal well-being).
Parental stress among intervention staff: Parental Stress Scale (PSS), total score | Pre-assessment and 6 - 8 weeks after pre-assessment
  The PSS is an 18-item self-report questionnaire. Items are rated on a 5-point Likert scale (1 = Strongly disagree, 2 = Disagree, 3 = Undecided, 4 = Agree, 5 = Strongly agree) and scores range from 18 to 90, with higher values indicating greater levels of parental stress.
Fidelity of intervention delivery: PLH-Facilitator Assessment Tool (PLH-FAT) | During the implementation of the intervention (6 - 8 weeks)
  The assessment tool focuses on various aspects of facilitator performance, and includes the percentage score on the completion of intervention activities and the percentage score on the demonstration of intervention skills.
Attendance rate - Other Subscales | During the implementation of the intervention (6 - 8 weeks)
  Percentage of group PLH sessions attended by both adolescent and caregiver in a given family (family attendance); Percentage of catch-up PLH contact out of 6 (family); Percentage of adolescents attending Magnificent Mei (1 session) and I Support My Friends (2 sessions).
Enrollment rate | During the implementation of the intervention (Six weeks)
  Percentage of participants who joined the study and have attended at least one group PLH session (individual enrollment for adolescents and caregivers) and percentage of families where both adolescent and caregiver attended at least one group PLH session (family enrollment).
Intervention costs | During the implementation of the intervention (6 - 8 weeks)
  Personnel time resources associated with the training and delivery of the intervention, organizational, material, transportation and consumable costs.
Adolescent defined problems: The Top Problem Assessment | Pre-assessment and 6 - 8 weeks after pre-assessment
  The Top Problem Assessment assesses adolescents' problems they are most concerned about. They can name three problems they choose and provide numerical severity ratings on a scale ranging from 0 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Foran, Prof, Principal Investigator — University of Klagenfurt; Yulia Shenderovich, Dr, Principal Investigator — Cardiff University; Marija Raleva, Prof, Principal Investigator — Institute for Marriage, Family and Systemic Practice - ALTERNATIVA; Galina Lesco, Dr., Principal Investigator — Health for Youth Association, Moldova; Graham Moore, Prof, Principal Investigator — Cardiff University; Rhiannon Evans, Prof, Principal Investigator — Cardiff University; Judit Simon, Prof, Principal Investigator — Medical University of Vienna; Nina Heinrichs, Prof, Principal Investigator — Bielefeld University; Nevena Calovska, Prof, Principal Investigator — Association of Systemic Therapists Education Centre; Bojan Shimbov, Prof, Principal Investigator — University Jaume I Castellon, Spain
Locations (1):
- Institute Alternativa, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: Yes
The project has a detailed data management plan (DMP) that defines data sharing procedures. The DMP was provided as a deliverable to the European Commission and is updated throughout the study funding period.
Supporting Information: Study Protocol
Time Frame: After completion of the study and publication of the main results.
Access Criteria: Prof. Heather Foran is responsible for data management of the FLOURISH project. For information related to data sharing, please contact her at heather.foran@aau.at
URL: https://www.flourish-study.org

REFERENCES:
- [Derived] Piolanti A, Mueller J, Waller F, Heinrichs N, Simon J, Shenderovich Y, Sampathkumar S, Wienand D, Raleva M, Kunovski I, Babii V, Zhao X, Moore G, Foran HM. Family-focused intervention programme to foster adolescent mental health and well-being: protocol for a multicountry cluster randomised factorial trial (FLOURISH Phase 2). BMJ Open. 2025 Feb 7;15(2):e094085. doi: 10.1136/bmjopen-2024-094085. PMID 39920046